CLINICAL TRIAL: NCT06515457
Title: A Clinical Trial to Evaluate the Efficacy of an Oral Supplement in Supporting Vision and Eye Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bio Nature Health (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20425
Record Dates: First submitted 2024-07-17; First posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Inflammation Symptoms; Eye Dryness; Eye Health
Keywords: Vision Health; Eye Empower
MeSH Terms: conditions — Xerophthalmia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Eye Empower Supplement Arm (Experimental): Participants in this arm will take three capsules of BioNatureHealth's Eye Empower supplement daily for three weeks.
  Interventions: Dietary Supplement: Eye Empower

INTERVENTIONS:
Dietary Supplement: Eye Empower — Participants will take three capsules of the Eye Empower supplement daily for three weeks.
  Other Names: BioNatureHealth Eye Empower

SUMMARY:
This study aims to evaluate the efficacy of BioNatureHealth's Eye Empower supplement in supporting vision and eye health. It is a virtual, single-group trial lasting 3 weeks. Participants will take three capsules of the supplement daily and complete questionnaires at Baseline, Week 1, Week 2, and Week 3 to assess visual clarity, dryness, symptoms of inflammation, and sensitivity to blue light.

ELIGIBILITY:
Inclusion Criteria:

* Male or female at birth, aged 40 or over
* Self-reported concerns about at least two of the following symptoms: dry eyes, red/itchy/irritated eyes, sensitivity to blue light, blurred vision (far or near)
* Generally healthy without uncontrolled chronic diseases
* Willing to avoid using new eye health prescriptions, over-the-counter medications, supplements, and herbal remedies for the study duration
* Consistent use of current eye health supplements or herbal remedies for at least 3 months prior to the study
* Willing to maintain current diet, sleep schedule, and activity level during the study

Exclusion Criteria:

* Pre-existing chronic conditions preventing protocol adherence, including oncological and psychiatric disorders
* Diagnosed diabetes (Type I or II)
* Planning to undergo any eye-related procedures during the study
* Recent surgeries or invasive treatments within the last six months
* History of major illness within the last three months
* Recent use of a supplement with active ingredients in the test product
* Severe allergic reactions requiring an EpiPen, including shellfish allergy
* Pregnant, breastfeeding, or planning to conceive
* Use of medications or herbal supplements that impact the blood
* Non-consumption of animal products for religious or personal reasons
* Unwillingness to follow the study protocol
* Anyone with a history of drug or alcohol abuse

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-04-22 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Improvement in Visual Clarity | Baseline, Week 1, Week 2, and Week 3
  Participants will report on their visual clarity through self-reported questionnaires. The questionnaires will evaluate changes in visual clarity from baseline.
Reduction in Eye Dryness | Baseline, Week 1, Week 2, Week 3
  Participants will self-report changes in eye dryness through questionnaires administered at specific intervals during the study. Parameters include the frequency and severity of dry eye symptoms.
Reduction in Symptoms of Inflammation | Baseline, Week 1, Week 2, Week 3
  Participants will self-report changes in symptoms of eye inflammation through questionnaires administered at specific intervals during the study. Parameters include redness, irritation, and discomfort.
Reduction in Sensitivity to Blue Light | Baseline, Week 1, Week 2, Week 3
  Participants will self-report changes in sensitivity to blue light through questionnaires administered at specific intervals during the study. Parameters include the degree of discomfort experienced when exposed to blue light from screens and other sources.

SECONDARY OUTCOMES:
Improvement in Overall Eye Health | Baseline, Week 1, Week 2, and Week 3
  Participants will report on their overall eye health through self-reported questionnaires. The questionnaires will assess changes in symptoms such as eye dryness, symptoms of inflammation, and sensitivity to blue light.

CONTACTS AND LOCATIONS:
Locations (1):
- Citruslabs, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: No